CLINICAL TRIAL: NCT00865215
Title: A Relative Bioavailability Study of 160 mg Propranolol Hydrochloride Extended Release Capsules Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of Propranolol Hydrochloride 160 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R05-1383
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Propranolol; Healthy subjects
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Propranolol Hydrochloride Extended Release Capsules 160 mg, single dose
  Interventions: Drug: Propranolol Hydrochloride Extended Release Capsules 160 mg
- B (Active Comparator): INDERAL® LA 160 mg Capsules, single dose
  Interventions: Drug: INDERAL® LA 160 mg Capsules, single dose

INTERVENTIONS:
Drug: Propranolol Hydrochloride Extended Release Capsules 160 mg — A: Experimental Subjects received Actavis formulated products under fasting conditions
  Other Names: Propranolol
  Arms: A
Drug: INDERAL® LA 160 mg Capsules, single dose — B: Active comparator Subjects received Wyeth Pharmaceuticals formulated products under fasting conditions
  Other Names: Propranolol
  Arms: B

SUMMARY:
The purpose of this study is TO compare the relative bioavailability of Propranolol Hydrochloride Extended Release Capsules 160 mg (Actavis) with that of INDERAL® LA 160 mg Capsules (Wyeth Pharmaceuticals) following a single oral dose (1 x 160 mg) in healthy adult volunteers under fasting conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, single dose, two-way crossover study under fasting conditions

Official Title: A Relative Bioavailability Study of 160 mg Propranolol Hydrochloride Extended Release Capsules Under Fasting Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers who have been informed of the nature of the study and agree to read, review and sign the informed consent document prior to Period I dosing.
2. Volunteers who have completed the screening process within 28 days prior to Period I dosing.
3. Volunteers who are healthy adult men and women 18 to 50 years of age, inclusive, at the time of dosing.
4. Volunteers who have a body mass index (BMI) between 18-32 kg/m2, inclusive, and weigh at least 110 lbs.
5. Volunteers who are healthy as documented by the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and by general observations. Any abnormalities/deviations from the normal range that might be considered clinically relevant by the study physician and investigator will be evaluated for individual cases, documented in study files, and agreed upon by both the study physician and investigator prior to enrolling the volunteer in this study and for continued enrollment.
6. Volunteers who have a negative urine drug screen.
7. Female volunteers must have a negative pregnancy screen.
8. Female volunteers practicing an acceptable method of birth control as judged by the investigator(s), such as condom with spermicide, diaphragm with spermicide, intrauterine device (IUD), or abstinence throughout the duration of the study; or of postmenopausal (no menses) status for at least 1 year; or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

1. Volunteers who report receiving any investigational drug within 28 days prior to Period I dosing.
2. Volunteers who report any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease as determined by the clinical investigator(s).
3. Volunteers whose clinical laboratory test values outside the accepted reference range and when confirmed on re-examination is deemed to be clinically significant.
4. Volunteers who demonstrate a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
5. Volunteers who report a history of allergic response(s) to propranolol or related drugs.
6. Volunteers who report the use of any systemic prescription medication in the 14 days prior to Period I dosing.
7. Volunteers who report the use of any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
8. Volunteers who report a history of clinically significant allergies including drug allergies.
9. Volunteers who report a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
10. Volunteers who report a history of drug or alcohol addiction or abuse within the past year.
11. Volunteers who demonstrate a positive drug abuse screen for this study prior to Period I dose administration.
12. Volunteers who currently use tobacco products.
13. Volunteers who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
14. Volunteers who report donating plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
15. Volunteers who demonstrate a positive pregnancy screen (females only).
16. Volunteers who are currently pregnant or breastfeeding (females only).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-04; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson,, Pharm.D,, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States